CLINICAL TRIAL: NCT01526785
Title: A Phase 4 Open Label, Prospective Study in Patients With Pompe Disease to Evaluate The Efficacy and Safety of Alglucosidase Alfa Produced at the 4000L Scale
Brief Title: A Study to Evaluate the Efficacy and Safety of Alglucosidase Alfa Produced at the 4000 L Scale for Pompe Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to approved label expansion
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU09411; EFC12720 (Other: Sanofi)
Record Dates: First submitted 2012-02-02; First posted 2012-02-06 (Estimated); Results first posted 2015-10-27 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alglucosidase alfa (Experimental): Alglucosidase alfa (4000 L scale) intravenous (IV) infusion administered for 52 weeks as per physician's routine practice.
  Interventions: Drug: Alglucosidase alfa

INTERVENTIONS:
Drug: Alglucosidase alfa — 4000 L alglucosidase alfa administered by IV infusion at the same dose and dose regimen used for the patient's routine treatment prior to the study for 52 weeks.
  Other Names: Lumizyme®

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of treatment with 4000 litre (L) alglucosidase alfa (Lumizyme®) in Pompe participants.

ELIGIBILITY:
Inclusion Criteria:

A participant might meet all of the following criteria to be eligible for this study.

1. The participant and/or their parent/legal guardian was willing and able to provide signed informed consent.
2. The participant might be at least 1 year of age at the time of informed consent.
3. The participant had a diagnosis of Pompe disease and might have received treatment with 160 L alglucosidase alfa prior to screening.
4. The participant, if female and of childbearing potential, might have a negative pregnancy test (urine beta-human chorionic gonadotropin) at baseline. Note: all female participants of childbearing potential and sexually mature males might agree to use a medically accepted method of contraception throughout the study.

Exclusion Criteria:

A participant who met any of the following criteria were to be excluded from this study.

1. The participant had within the past 3 months received or was currently receiving any investigational product other than 160 L alglucosidase alfa or was currently participating in another clinical treatment study.
2. The participant, in the opinion of the Investigator, was clinically unstable and would not be expected to survive to completion of the 52-week treatment period.
3. The participant and/or their parent/legal guardian, in the opinion of the Investigator, was unable to adhere to the requirements of the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (51):
- United States (51):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Oakland, California
  - Orange, California
  - San Diego, California
  - San Jose, California
  - Stanford, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - Glens Falls, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Valhalla, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Miliwaukee, Wisconsin

REFERENCES:
- [Derived] Duong T, Kishnani PS, An Haack K, Foster MC, Gibson JB, Wilson C, Hahn SH, Hillman R, Kronn D, Leslie ND, Pena LDM, Sparks SE, Stockton DW, Tanpaiboon P, Day JW; Pompe ADVANCE Study Consortium. Motor Responses in Pediatric Pompe Disease in the ADVANCE Participant Cohort. J Neuromuscul Dis. 2022;9(6):713-730. doi: 10.3233/JND-210784. PMID 36214004
- [Derived] Byrne BJ, Colan SD, Kishnani PS, Foster MC, Sparks SE, Gibson JB, An Haack K, Stockton DW, Pena LDM, Hahn SH, Johnson J, Tanpaiboon PX, Leslie ND, Kronn D, Hillman RE, Wang RY; Pompe ADVANCE Study Consortium. Cardiac responses in paediatric Pompe disease in the ADVANCE patient cohort. Cardiol Young. 2022 Mar;32(3):364-373. doi: 10.1017/S1047951121002079. Epub 2021 Aug 23. PMID 34420548
- [Derived] Kishnani PS, Gibson JB, Gambello MJ, Hillman R, Stockton DW, Kronn D, Leslie ND, Pena LDM, Tanpaiboon P, Day JW, Wang RY, Goldstein JL, An Haack K, Sparks SE, Zhao Y, Hahn SH; Pompe ADVANCE Study Consortium. Clinical characteristics and genotypes in the ADVANCE baseline data set, a comprehensive cohort of US children and adolescents with Pompe disease. Genet Med. 2019 Nov;21(11):2543-2551. doi: 10.1038/s41436-019-0527-9. Epub 2019 May 14. PMID 31086307
- [Derived] Hahn SH, Kronn D, Leslie ND, Pena LDM, Tanpaiboon P, Gambello MJ, Gibson JB, Hillman R, Stockton DW, Day JW, Wang RY, An Haack K, Shafi R, Sparks S, Zhao Y, Wilson C, Kishnani PS; Pompe ADVANCE Study Consortium. Efficacy, safety profile, and immunogenicity of alglucosidase alfa produced at the 4,000-liter scale in US children and adolescents with Pompe disease: ADVANCE, a phase IV, open-label, prospective study. Genet Med. 2018 Oct;20(10):1284-1294. doi: 10.1038/gim.2018.2. Epub 2018 Mar 22. PMID 29565424

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in the United States. A total of 113 participants were treated between 9 March 2012 and 4 June 2014.
Groups:
- Alglucosidase Alfa: Alglucosidase alfa (4000 litre [L] scale) intravenous (IV) infusion administered for 52 weeks as per physician's routine practice.
Period: Overall Study
Arm/Group | Alglucosidase Alfa
Started | 113
Completed | 100
Not Completed | 13
Not completed — Study Terminated by Sponsor | 8
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Full analysis population defined as all participants who receive at least 1 infusion of 4000 L alglucosidase alfa during the study.
Groups:
- Alglucosidase Alfa: Alglucosidase alfa (4000 L scale) IV infusion administered for 52 weeks as per physician's routine practice.
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.8 (3.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Clinically Stable or Improved at Week 52
Description: Clinical stability was defined as absence of death due to disease progression or new dependency on invasive ventilation and; decline in cardiac status, motor function, and pulmonary function from baseline.
Time Frame: Week 52
Population: Full analysis population. Number of participants analyzed = participants with available data at Week 52 for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 104
percentage of participants | 83.7 [75.1 to 90.2]

2. Secondary Outcome: Survival Rate at Week 52
Description: Percentage of participants who were alive at Week 52, were reported. Survival rate was calculated by Kaplan-Meier estimate.
Time Frame: Week 52
Population: Full analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 113
percentage of participants | 98.1 [92.73 to 99.53]

3. Secondary Outcome: Invasive Ventilator-Free Survival Rate at Week 52
Description: Percentage of participants, who were invasive ventilator-free at week 52, are reported. Invasive ventilation was defined as mechanical ventilatory support applied with the use of an endotracheal tube or tracheostomy. Invasive ventilator-free survival rate was calculated by Kaplan-Meier estimate.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 81
percentage of participants | 92.4 [83.89 to 96.53]

4. Secondary Outcome: Change From Baseline on Left Ventricular Mass Z-Score (LVM-Z) at Week 52
Description: Z-Scores indicate the number of standard deviations (SD) from the mean in a normal distribution. A negative change from baseline indicates an increase in LVM-Z score. The normal range is -2 to 2 and greater than 2 may indicate left ventricular hypertrophy.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 67
Z score | -0.5 (1.71)

5. Secondary Outcome: Change From Baseline on Gross Motor Function Measure-88 (GMFM-88) at Week 52
Description: GMFM-88 (88-item measure to detect gross motor function) consists of 5 components, each measured on a 4-point Likert scale.The score for each dimension was expressed as a percentage of the maximum score for that dimension.Total score ranges from 0% to 100%, where higher scores indicate better motor functions.
Time Frame: Baseline, Week 52
Population: Full analysis population. Number of participants analysed = participants with baseline and Week 52 GMFM-88 data.
Measure: Mean (Standard Deviation); unit: percentage of total score
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 90
percentage of total score | 3.7 (17.46)

6. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Week 52- At Supine Position
Description: Percent predicted FVC values are reported. FVC is the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in litres. Predicted forced vital capacity is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%.
Time Frame: Baseline, Week 52
Population: Full analysis population. Number of participants analysed = participants with baseline and Week 52 FVC data.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 13
percent predicted FVC | 3.2 (11.07)

7. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Week 52- At Sitting Position
Description: as for outcome 6
Time Frame: Baseline, Week 52
Population: Full analysis population. Number of participants analysed = participants with baseline and Week 52 FVC data.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Alglucosidase Alfa
Number analyzed (Participants) | 22
percent predicted FVC | 2.3 (11.8)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 52) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the first infusion of study drug up to 30 days after last infusion of study drug). Analysis was performed on safety population which included all treated participants.
Groups:
- Alglucosidase Alfa: Alglucosidase alfa (4000 L scale) IV infusion administered for 52 weeks as per participant's routine practice.
Arm/Group | Alglucosidase Alfa
Serious Adverse Events (participants affected / at risk) | 73/113
Other Adverse Events (participants affected / at risk) | 113/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa (N=113)
Bradycardia (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 3
Cardiopulmonary failure (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Left ventricular hypertrophy (Cardiac disorders) | 2
Mitral valve incompetence (Cardiac disorders) | 1
Pulseless electrical activity (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 4
Tachycardia (Cardiac disorders) | 1
Motion sickness (Ear and labyrinth disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 2
Chills (General disorders) | 2
Device breakage (General disorders) | 1
Device malfunction (General disorders) | 1
Hypothermia (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 10
Cholecystitis acute (Hepatobiliary disorders) | 1
Adenovirus infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Bacterial tracheitis (Infections and infestations) | 2
Bronchiolitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 3
Haemophilus bacteraemia (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Klebsiella bacteraemia (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Metapneumovirus infection (Infections and infestations) | 3
Otitis media acute (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Periumbilical abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 25
Pneumonia parainfluenzae viral (Infections and infestations) | 1
Pneumonia pseudomonal (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 2
Pneumonia viral (Infections and infestations) | 3
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 4
Respiratory tract infection viral (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 5
Tracheostomy infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Urinary tract infection bacterial (Infections and infestations) | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Feeding tube complication (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Oxygen saturation decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Failure to thrive (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Brain injury (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Gross motor delay (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Self-injurious ideation (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 16
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Central venous catheterisation (Surgical and medical procedures) | 1
Therapeutic procedure (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa (N=113)
Anaemia (Blood and lymphatic system disorders) | 7
Coagulopathy (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 2
Bundle branch block right (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Defect conduction intraventricular (Cardiac disorders) | 4
Diastolic dysfunction (Cardiac disorders) | 1
Heart valve incompetence (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 5
Right atrial dilatation (Cardiac disorders) | 1
Right ventricular hypertrophy (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 13
Tricuspid valve incompetence (Cardiac disorders) | 1
Wolff-Parkinson-White syndrome (Cardiac disorders) | 2
Cryptorchism (Congenital, familial and genetic disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 3
Conductive deafness (Ear and labyrinth disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 5
Eustachian tube dysfunction (Ear and labyrinth disorders) | 5
Middle ear effusion (Ear and labyrinth disorders) | 5
Mixed deafness (Ear and labyrinth disorders) | 1
Otorrhoea (Ear and labyrinth disorders) | 3
Tympanic membrane disorder (Ear and labyrinth disorders) | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Precocious puberty (Endocrine disorders) | 2
Astigmatism (Eye disorders) | 2
Blepharitis (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Dry eye (Eye disorders) | 4
Eye discharge (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 4
Hypermetropia (Eye disorders) | 1
Lid sulcus deepened (Eye disorders) | 1
Myopia (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Strabismus (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 10
Abdominal pain upper (Gastrointestinal disorders) | 11
Abnormal faeces (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 20
Dental caries (Gastrointestinal disorders) | 3
Dental discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 55
Dysphagia (Gastrointestinal disorders) | 2
Faecal incontinence (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Gingival bleeding (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Infrequent bowel movements (Gastrointestinal disorders) | 1
Lip blister (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 12
Oral disorder (Gastrointestinal disorders) | 1
Rectal fissure (Gastrointestinal disorders) | 1
Regurgitation (Gastrointestinal disorders) | 1
Retained deciduous tooth (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 2
Sensitivity of teeth (Gastrointestinal disorders) | 1
Teething (Gastrointestinal disorders) | 4
Tongue spasm (Gastrointestinal disorders) | 1
Tooth deposit (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 42
Abasia (General disorders) | 1
Asthenia (General disorders) | 4
Catheter site erythema (General disorders) | 1
Catheter site extravasation (General disorders) | 4
Catheter site haemorrhage (General disorders) | 1
Catheter site inflammation (General disorders) | 1
Catheter site oedema (General disorders) | 1
Catheter site pain (General disorders) | 3
Catheter site rash (General disorders) | 1
Catheter site related reaction (General disorders) | 1
Catheter site swelling (General disorders) | 1
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 6
Chills (General disorders) | 2
Crepitations (General disorders) | 1
Device breakage (General disorders) | 1
Device dislocation (General disorders) | 4
Device issue (General disorders) | 1
Device malfunction (General disorders) | 9
Device occlusion (General disorders) | 13
Discomfort (General disorders) | 2
Disease progression (General disorders) | 1
Energy increased (General disorders) | 1
Extravasation (General disorders) | 2
Fatigue (General disorders) | 4
Feeling hot (General disorders) | 1
Gait disturbance (General disorders) | 1
Granuloma (General disorders) | 2
Gravitational oedema (General disorders) | 1
Influenza like illness (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Infusion site swelling (General disorders) | 2
Injection site extravasation (General disorders) | 1
Injection site swelling (General disorders) | 1
Malaise (General disorders) | 2
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 3
Peripheral swelling (General disorders) | 4
Pyrexia (General disorders) | 61
Secretion discharge (General disorders) | 6
Thirst (General disorders) | 1
Thrombosis in device (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic fibrosis (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Food allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 5
Multiple allergies (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Abscess limb (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Adenovirus infection (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacterial tracheitis (Infections and infestations) | 5
Beta haemolytic streptococcal infection (Infections and infestations) | 1
Body tinea (Infections and infestations) | 3
Bronchiolitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 8
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 7
Croup infectious (Infections and infestations) | 2
Device related infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 12
Ear lobe infection (Infections and infestations) | 1
Enterovirus infection (Infections and infestations) | 1
Erythema infectiosum (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 11
Gastroenteritis norovirus (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 4
Gastrointestinal infection (Infections and infestations) | 1
Gingival abscess (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 3
Impetigo (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 8
Labyrinthitis (Infections and infestations) | 1
Lice infestation (Infections and infestations) | 1
Lip infection (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 12
Oral candidiasis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 2
Otitis externa fungal (Infections and infestations) | 1
Otitis media (Infections and infestations) | 23
Otitis media acute (Infections and infestations) | 6
Otitis media chronic (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 7
Pharyngitis streptococcal (Infections and infestations) | 13
Pneumonia (Infections and infestations) | 17
Pneumonia viral (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 4
Rash pustular (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 6
Rhinovirus infection (Infections and infestations) | 3
Rotavirus infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 5
Skin infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 3
Stoma site infection (Infections and infestations) | 2
Streptococcal infection (Infections and infestations) | 2
Streptococcal urinary tract infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 7
Tracheobronchitis (Infections and infestations) | 1
Tracheostomy infection (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 49
Upper respiratory tract infection bacterial (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 19
Viral infection (Infections and infestations) | 15
Viral rash (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 5
Vulvovaginal mycotic infection (Infections and infestations) | 1
Agitation postoperative (Injury, poisoning and procedural complications) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Animal scratch (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 7
Arthropod sting (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 6
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1
Eye contusion (Injury, poisoning and procedural complications) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 11
Feeding tube complication (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 2
Foreign body (Injury, poisoning and procedural complications) | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 6
Laryngeal injury (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 5
Limb injury (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Postoperative fever (Injury, poisoning and procedural complications) | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 8
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 9
Skin wound (Injury, poisoning and procedural complications) | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1
Splinter (Injury, poisoning and procedural complications) | 1
Stoma site erythema (Injury, poisoning and procedural complications) | 2
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 2
Stoma site irritation (Injury, poisoning and procedural complications) | 3
Stoma site rash (Injury, poisoning and procedural complications) | 1
Stoma site reaction (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1
Tooth avulsion (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Tooth injury (Injury, poisoning and procedural complications) | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 2
Vaccination complication (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase abnormal (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase abnormal (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 4
Atrial pressure increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatine phosphokinase MB increased (Investigations) | 7
Blood creatine phosphokinase abnormal (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 7
Blood culture positive (Investigations) | 1
Blood lactate dehydrogenase abnormal (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Blood potassium decreased (Investigations) | 2
Blood pressure decreased (Investigations) | 2
Blood pressure increased (Investigations) | 7
Blood pressure systolic increased (Investigations) | 1
Blood uric acid decreased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Blood zinc decreased (Investigations) | 1
Body temperature increased (Investigations) | 5
Brain natriuretic peptide increased (Investigations) | 5
Breath sounds abnormal (Investigations) | 2
Creatine urine increased (Investigations) | 1
Creatinine urine increased (Investigations) | 1
Electrocardiogram PR shortened (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Electrocardiogram ST segment elevation (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 2
Eosinophil count increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 3
Heart rate increased (Investigations) | 5
Liver function test abnormal (Investigations) | 1
Neutrophil count abnormal (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Neutrophil percentage increased (Investigations) | 1
Occult blood positive (Investigations) | 1
Oxygen saturation decreased (Investigations) | 4
Platelet count increased (Investigations) | 2
Protein urine (Investigations) | 1
Protein urine present (Investigations) | 1
Pulmonary function test decreased (Investigations) | 2
Pulse pressure abnormal (Investigations) | 1
Respiratory rate increased (Investigations) | 1
Serum ferritin decreased (Investigations) | 1
Specific gravity urine (Investigations) | 1
Sputum culture positive (Investigations) | 1
Staphylococcus test positive (Investigations) | 1
Tuberculin test positive (Investigations) | 1
Urine ketone body present (Investigations) | 1
Urine output decreased (Investigations) | 2
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 3
White blood cell count abnormal (Investigations) | 1
White blood cell count increased (Investigations) | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 5
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2
Iron deficiency (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Deformity thorax (Musculoskeletal and connective tissue disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2
Fracture pain (Musculoskeletal and connective tissue disorders) | 1
Hip deformity (Musculoskeletal and connective tissue disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Kyphosis (Musculoskeletal and connective tissue disorders) | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 6
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 2
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 3
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Allodynia (Nervous system disorders) | 1
Areflexia (Nervous system disorders) | 2
Burning sensation (Nervous system disorders) | 1
Clumsiness (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Facial paresis (Nervous system disorders) | 1
Formication (Nervous system disorders) | 1
Gross motor delay (Nervous system disorders) | 2
Headache (Nervous system disorders) | 14
Hypoaesthesia (Nervous system disorders) | 1
Hyporeflexia (Nervous system disorders) | 2
Hypotonia (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 4
Motor developmental delay (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 2
Muscle contractions involuntary (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paralysis flaccid (Nervous system disorders) | 1
Poor quality sleep (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 5
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 2
Bruxism (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 1
Oppositional defiant disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 4
Urinary retention (Renal and urinary disorders) | 1
Genital discomfort (Reproductive system and breast disorders) | 2
Vaginal prolapse (Reproductive system and breast disorders) | 1
Vulvovaginal disorder (Reproductive system and breast disorders) | 1
Vulvovaginal erythema (Reproductive system and breast disorders) | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 5
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 7
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 8
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 7
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 24
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Snoring (Respiratory, thoracic and mediastinal disorders) | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2
Tracheal ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 8
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 5
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 4
Granuloma skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1
Macule (Skin and subcutaneous tissue disorders) | 2
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 31
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Red man syndrome (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 9
Central venous catheterisation (Surgical and medical procedures) | 1
Ear tube removal (Surgical and medical procedures) | 1
Gastrostomy tube removal (Surgical and medical procedures) | 1
Aortic dilatation (Vascular disorders) | 1
Flushing (Vascular disorders) | 7
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 2
Pallor (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.